CLINICAL TRIAL: NCT00732303
Title: A Phase II Study of Concurrent Pemetrexed and Radiation for Poor-Risk Stage III Non-Small Cell Lung Cancer: Hoosier Oncology Group LUN08-129
Brief Title: Pemetrexed and Radiation for Poor-Risk Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to withdrawal of pharmaceutical funding
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN08-129
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Results first posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): * Pemetrexed (Alimta) 500mg/m^2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  * Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
  Interventions: Drug: Pemetrexed; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed (Alimta) 500mg/^2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
Radiation: Radiation Therapy — Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.

SUMMARY:
Pemetrexed is approved for second line therapy in metastatic NSCLC. Given the single-agent activity of pemetrexed and the tolerability of pemetrexed in combination with radiation, this study will evaluate survival rates and toxicities in patients with poor risk stage III NSCLC.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Pemetrexed (Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
* Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.

The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.

Performance Status: ECOG performance status 2

Life Expectancy: Not specified

Hematopoietic:

* Platelets ≥ 100 K/mm3
* Absolute Neutrophil Count (ANC) ≥ 2.0 K/mm3

Hepatic:

* Aspartate transaminase (AST) ≤ 2.5 x ULN.
* Alanine transaminase (ALT) ≤ 2.5 x ULN.
* Total bilirubin ≤ 1.5 x ULN

Renal:

* Calculated creatinine clearance (using Cockcroft-Gault formula) ≥ 45 cc/min

Cardiovascular:

* No significant history of cardiac disease. Must not have unstable angina (anginal symptoms at rest).

Pulmonary:

* Forced expiratory volume in 1 second (FEV1) greater than 1L

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of Non Small Cell Lung Cancer (NSCLC)
* Measurable or non-measurable disease per RECIST as evaluated by imaging within 28 days prior to registration for protocol therapy
* Unresectable Stage IIIA or IIIB disease as evaluated by imaging within 28 days prior to registration for protocol therapy
* Weight loss of greater than 10% in the preceding six months prior to registration for protocol therapy.
* Serum albumin < 0.85 x institutional lower limit of normal
* Able and willing to interrupt non-steroidal anti-inflammatory agents for 2 days before (5 days for long acting agents such as piroxicam), the day of, and 2 days following administration of pemetrexed
* Lung V20 < 35% within 14 days prior to registration for protocol therapy, as planned by the radiation oncologist
* Mean lung dose < 20 Gy within 14 days prior to registration for protocol therapy, as planned by the radiation oncologist
* Written informed consent and HIPAA authorization for release of personal health information
* Age ≥ 18 years
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time of consent until at least 90 days following completion of study treatment.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to registration for protocol therapy. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.

Exclusion Criteria:

* Patients with malignant pleural effusions are not eligible. The only exception is a patient with a pleural effusion visible only on CT scan (and not visible on CXR) OR deemed too small to tap.• No CNS metastases. All patients must undergo a CT scan/MRI of the brain within 28 days prior to registration for protocol therapy to exclude brain metastasis.
* No prior chemotherapy, adjuvant therapy or radiotherapy for lung cancer.
* No metastatic disease as determined by PET scan within 28 days prior to registration for protocol therapy.
* No active clinically serious infections as judged by the treating investigator (> CTC v3, Grade 2) including known human immunodeficiency virus (HIV) infection or chronic Hepatitis B or C.
* No other active malignancies.
* No history of collagen vascular disease (CVD).
* No significant history of cardiac disease. Must not have unstable angina (anginal symptoms at rest).
* No history of psychiatric illness/social situations that would limit compliance with study requirements.
* Females must not be breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Cancer Research Network
Locations (18):
- United States (18):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - NorthShore University Health System - Kellogg Cancer Center, Evanston, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - IN Onc/Hem Associates, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Hematology Oncology Associates S.J., P.A., Mount Holly, New Jersey
  - Providence Portland Medical Center, Portland, Oregon
  - Pennsylvania Oncology-Hematology Associates, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center Extramural Research Program, Rockledge, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Assignment: * Pemetrexed (Alimta) 500mg/m^2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x3 cycles
  * Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
  Pemetrexed: Pemetrexed(Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  Radiation Therapy:
  Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
Period: Overall Study
Arm/Group | Single Arm Assignment
Started | 8
Completed | 6
Not Completed | 2
Not completed — Study Terminated | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Assignment: * Pemetrexed (Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  * Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
  Pemetrexed: Pemetrexed(Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  Radiation Therapy:
  Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 68.50 [56 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To determine progression free survival in patients with poor risk stage III NSCLC treated with pemetrexed and concurrent definitive radiation
Time Frame: 24 months
Population: No data was collected and analyzed for this outcome measure due to termination of the study
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess Safety and Toxicity
Description: - To determine the toxicities of pemetrexed and concurrent definitive radiation in patients with poor risk stage III NSCLC.
Time Frame: 24 months
Population: Most frequent toxicities reported.
Measure: Number; unit: participants
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 8
participants
  Grade 1 and Grade 2 Fatigue | 7
  Grade 1 and 2 Anorexia | 6
  Grade 1 and 2 Cough | 6
  Grade 3 and 4 Fatigue | 4
  Grade 3 and 4 Anorexia | 3
  Grade 3 and 4 Neutropenia | 3

3. Secondary Outcome: Overall Survival
Description: To determine overall survival of pemetrexed and concurrent definitive radiation in patients with poor risk stage III NSCLC.
Time Frame: 24 months
Population: No data was collected and analyzed for this outcome measure due to termination of the study.
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting at baseline screening until participants went off treatment, which was a maximum of three cycles (months)
Groups:
- Pemetrexed\Radiation: * Pemetrexed (Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  * Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
  Pemetrexed: Pemetrexed(Alimta) 500mg/m2 administered intravenously over approximately 10-minutes on Day 1 of a 21-day cycle x 3 cycles
  Radiation Therapy:
  Radiation will start between days -1 to 2 from day 1 of cycle 1. Day 1 radiotherapy must be a Monday, Tuesday, or Wednesday.
  The planned radiation dose is 60 Gy in 2.0 Gy fractions. The entire PTV, including primary tumor and areas of known nodal disease, shall receive 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks.
Arm/Group | Pemetrexed\Radiation
Serious Adverse Events (participants affected / at risk) | 3/8
Other Adverse Events (participants affected / at risk) | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed\Radiation (N=8)
ANOREXIA (Gastrointestinal disorders) | 2 (2)
DEHYDRATION (Gastrointestinal disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed\Radiation (N=8)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 2 (9)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 6 (11)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (1)
CARDIAC ARRHYTHMIA (Cardiac disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 6 (7)
DEHYDRATION (Gastrointestinal disorders) | 2 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 3 (5)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 6 (18)
EDEMA: LIMB (Blood and lymphatic system disorders) | 2 (2)
ESOPHAGITIS (Gastrointestinal disorders) | 3 (4)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 6 (20)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 2 (2)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 2 (2)
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 (7)
HYPERTENSION (Cardiac disorders) | 1 (1)
HYPOTENSION (Cardiac disorders) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 4 (5)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 2 (5)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (7)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 3 (3)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 3 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 2 (3)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ESOPHAGUS (Gastrointestinal disorders) | 1 (3)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 4 (8)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 2 (5)
PAIN / BACK (General disorders) | 1 (1)
PAIN / CARDIAC/HEART (Cardiac disorders) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN - OTHER (General disorders) | 1 (1)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (6)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / RADIATION (Skin and subcutaneous tissue disorders) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 2 (5)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 2 (2)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (6)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No